CLINICAL TRIAL: NCT01031953
Title: Pilot Study of Fosaprepitant (MK-0517) for Breakthrough Chemotherapy Induced Nausea and Vomiting
Brief Title: Fosaprepitant Dimeglumine in Treating Patients With Nausea and Vomiting Caused By Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug contract timelines and inadequate enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joseph Bubalo, PharmD, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000612580; P30CA069533 (NIH); OHSU-HEM-08053-L (Other: OHSU 4498); NCT00939302 (obsolete NCT alias)
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Breakthrough Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Vomiting; Nausea | interventions — fosaprepitant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fosaprepitant (Experimental)
  Interventions: Drug: fosaprepitant dimeglumine; Drug: systemic chemotherapy; Other: survey administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: fosaprepitant dimeglumine — A 150 mg dose will be given to study patients as rescue therapy after chemotherapy only in the event of breakthrough nausea or vomiting.
Drug: systemic chemotherapy — Patients will receive chemotherapy on Day 1 of their scheduled therapeutic regimen in combination with the pre-defined standard 5-Hydroxytryptamine-3 (5HT3) antagonist, corticosteroid regimen, with or without benzodiazepine based on published guidelines3 or as clinically indicated
Other: survey administration — Prior to the first dose of chemotherapy patients will be instructed on how to complete their patient diary
Procedure: quality-of-life assessment — Patients will also be provided the Functional Living Index - Emesis (FLIE) quality of life survey to be completed at time zero and then after 24 hours

SUMMARY:
RATIONALE: Antiemetic drugs, such as fosaprepitant dimeglumine, may help lessen or prevent nausea and vomiting in patients treated with chemotherapy.

PURPOSE: This clinical trial is studying the side effects of fosaprepitant dimeglumine and to see how well it works in treating patients with nausea and vomiting caused by chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy and safety of fosaprepitant dimeglumine in patients with breakthrough chemotherapy-induced nausea and vomiting (CINV) after failing prophylactic antiemetic therapy.

Secondary

* To evaluate toxicity and serious adverse events associated with this regimen in these patients.
* To evaluate the ability of patients to tolerate oral intake.
* To evaluate the health-related quality of life of patients treated with this regimen.
* To evaluate specific side effects associated with this regimen, including pain sensation and/or soreness at the infusion site, headache, dizziness, and somnolence, in these patients .
* To refine the study design for future phase II and III studies of rescue therapy for breakthrough CINV using various secondary endpoints.

OUTLINE: Patients receive chemotherapy in combination with a pre-defined standard 5-Hydroxytryptamine-3 (5-HT3) antagonist or corticosteroid regimen with or without a benzodiazepine on day 1. If breakthrough nausea or vomiting occurs, patients then receive fosaprepitant dimeglumine IV once per standard administration guidelines. Patients with treatment response may receive additional doses of oral aprepitant once on days 2 and 3. Patients with persistent nausea/vomiting after 2 hours and who desire further treatment may receive standard rescue therapy with prochlorperazine, metoclopramide, or haloperidol with or without additional lorazepam until relief, at the discretion of the provider.

Patients complete a diary at baseline, and then at 2, 12, and 24 hours that includes a Visual Analogue Scale (VAS) for nausea; VAS for sedation; and questions about emesis and retching frequency, headache, dizziness, somnolence, and ability to take food and liquids orally. Patients also complete the Functional Living Index-Emesis Quality of Life survey at baseline and at 24 hours.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Scheduled to receive inpatient chemotherapy containing at least moderately emetogenic agents

  * May be given for adjuvant, neoadjuvant, curative, or palliative intent
  * May be given orally, IV, or by continuous infusion on ≥ 1 day
* Scheduled to receive 5-HT3 receptor antagonist antiemetic (e.g., ondansetron, granisetron, palonosetron, dolasetron mesylate, or dexamethasone with or without a benzodiazepine) on the day of chemotherapy
* Self-report of at least mild nausea (for which the patient feels needs rescuing) or moderate nausea (a score of ≥ 2 on a 4-point Likert scale) OR has had ≥ 1 episode of emesis since receiving chemotherapy
* No history of chronic nausea and/or vomiting (without chemotherapy), anticipatory nausea and/or vomiting, or emesis within 24 hours before chemotherapy
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* Able to understand English
* Not pregnant or nursing
* Negative pregnancy test
* No clinical evidence of current or impending bowel obstruction (i.e., tumor pressing on the bowel)
* No allergy or intolerance to study drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior chemotherapy allowed
* No aprepitant as prophylaxis or rescue treatment during the current course of chemotherapy (other than as a part of study therapy)
* Not scheduled to receive a dopamine antagonist after chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, PharmD, BCPS, BCOP, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from August 2008 until January 2013
Pre-assignment Details: There were 34 participants who signed the informed consent for this study but of these, only 11 received the study treatment. The other 23 were screen failures.
Groups:
- Fosaprepitant: A 150mg dose of study drug given to participants who experience breakthrough nausea and vomiting after prophylactic anti emetics given with chemotherapy
Period: Overall Study
Arm/Group | Fosaprepitant
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fosaprepitant
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Nausea Score From Baseline to 2 Hours as Assessed by the Numerical Visual Analogue Scale
Description: The outcome measure is the number of participants that self report improvement in a nausea score from baseline, prior to fosaprepitant, to 2 hours post dose. This includes only participants who report breakthrough nausea or vomiting after chemotherapy and after receiving prophylactic anti-emetics. The primary outcome is measured using the visual analogue scale, a self report scale from "No Nausea" to "Nausea as bad as it can be"; a value can be indicated anywhere on this scale using a free hand mark by the participant and gauged with ruler by study staff. Any participant that reported a lower value on the scale 2 hours from baseline would be considered in this outcome measure.
Time Frame: Baseline to 2 hours after study drug administered.
Measure: Number; unit: participants
Groups:
- Participants Receiving Fosaprepitant: A 150mg dose of study drug given to participants who experience breakthrough nausea and vomiting after prophylactic anti emetics given with chemotherapy
Arm/Group | Participants Receiving Fosaprepitant
Number analyzed (Participants) | 11
participants | 10

2. Secondary Outcome: Improvement in Nausea Score From Baseline to 12 Hours
Description: The outcome measure is the number of participants that self report improvement in a nausea score from baseline, prior to fosaprepitant, to 12 hours post dose. This includes only participants who report breakthrough nausea or vomiting after chemotherapy and after receiving prophylactic anti-emetics. The primary outcome is measured using the visual analogue scale, a self report scale from "No Nausea" to "Nausea as bad as it can be"; a value can be indicated anywhere on this scale using a free hand mark by the participant and gauged with ruler by study staff. Any participant that reported a lower value on the scale 12 hours from baseline would be considered in this outcome measure.
Time Frame: Baseline to 12 hours after study drug administered.
Measure: Number; unit: participants
Arm/Group | Participants Receiving Fosaprepitant
Number analyzed (Participants) | 11
participants | 11

3. Secondary Outcome: Improvement in Nausea Score From 2 Hours to 24 Hours
Description: The outcome measure is the number of participants that self report improvement in a nausea score from 2 hours after receiving fosaprepitant to 24 hours post dose. This includes only participants who report breakthrough nausea or vomiting after chemotherapy and after receiving prophylactic anti-emetics. The outcome is measured using the visual analogue scale, a self report scale from "No Nausea" to "Nausea as bad as it can be"; a value can be indicated anywhere on this scale using a free hand mark by the participant and gauged with ruler by study staff. Any participant reporting a lower value on the scale at the 12 or 24 hour time point would be considered in this outcome measure.
Time Frame: 2 hours to 24 hours after study drug administered.
Measure: Number; unit: participants
Groups:
- Change in Nausea Score From 2 Hours to 12 and 24 Hours: A 150mg dose of study drug given to participants who experience breakthrough nausea and vomiting after prophylactic anti emetics given with chemotherapy
Arm/Group | Change in Nausea Score From 2 Hours to 12 and 24 Hours
Number analyzed (Participants) | 11
participants | 7

4. Secondary Outcome: Number of Participants Who Experienced Vomiting Episodes From Baseline to 24 Hours
Description: Participants were asked to report any episodes of vomiting before (baseline) and up to 24 hours after receiving Fosaprepitant. The outcome considers the number of participants reporting any episodes of emesis after receiving Fosaprepitant.
Time Frame: Baseline to 24 hours after study drug administered.
Measure: Number; unit: participants
Groups:
- Participants Who Recieved Fosaprepitant: Number of participants who experienced vomiting episodes from baseline to 24 hours after receiving Fosaprepitant
Arm/Group | Participants Who Recieved Fosaprepitant
Number analyzed (Participants) | 11
participants | 2

5. Secondary Outcome: Participants Who Required the Use of Second Rescue Drug (Time to Treatment Failure)
Description: Participants with persistent nausea/vomiting after 2 hours and who desired further treatment, received standard rescue therapy at the discretion of provider with prochlorperazine, metoclopramide or haloperidol with or without additional lorazepam until relief
Time Frame: 2 hours after administration of Fosaprepitant 150 mg IV
Measure: Number; unit: participants
Groups:
- Participants That Received Fosaprepitant: This arm includes only those participants that required the use of second rescue drug after receiving Fosaprepitant
Arm/Group | Participants That Received Fosaprepitant
Number analyzed (Participants) | 11
participants | 9

6. Secondary Outcome: Participants Achieving a Complete Response (no Emesis, no Additional Rescue Medication Required)
Description: The recommended dose Fosaprepitant (MK-0517) is 115 mg administered intravenously 30 minutes before chemotherapy treatment. In this study, a 150 mg dose will be given to study patients as rescue therapy after chemotherapy only in the event of breakthrough nausea or vomiting. Those participants who did not report episodes of emesis or did not require additional rescue medications are measured in this outcome
Time Frame: up to 24 hours after receiving fosaprepitant
Measure: Number; unit: participants
Groups:
- Participants That Received Fosaprepitant: Number of participants achieving a Complete Response (CR) up to 24 hours after receiving fosaprepitant
Arm/Group | Participants That Received Fosaprepitant
Number analyzed (Participants) | 11
participants | 1

7. Secondary Outcome: Participants With Increased Fatigue or Sedation Within 24 Hours After Receiving Fosaprepitant
Description: Participants meeting this outcome self report experiencing drowsiness at any of the study time points (2, 12 or 24 hours after receiving fosaprepitant).
Time Frame: up to 24 hours after study drug administered.
Measure: Number; unit: participants
Groups:
- Participants That Received Fosaprepitant: participants with self report fatigue or sedation after receiving fosaprepitant
Arm/Group | Participants That Received Fosaprepitant
Number analyzed (Participants) | 11
participants | 7

8. Secondary Outcome: Participants With Specific Side Effects, Including Pain Sensation/Soreness at the Infusion Site, Headache, and Dizziness
Description: Participants who self report pain/soreness at drug infusion site, headache, or dizziness at any of the study time points (2, 12, or 24 hours after receiving fosaprepitant) are measured in this outcome.
Time Frame: up to 24 hours after study drug administered.
Measure: Number; unit: participants
Groups:
- Participants That Received Fosaprepitant: Only those in the study arm above that self report headache, dizziness, or pain/soreness at the infusion site are considered in this outcome
Arm/Group | Participants That Received Fosaprepitant
Number analyzed (Participants) | 11
participants | 5

ADVERSE EVENTS:
Arm/Group | Fosaprepitant
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant (N=11)
Dizziness (Nervous system disorders) | 1 (1)
Confusion-ifosfamide encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
* Missing data did affect results for the 24 hour mark
* Lack of control group to measure possible neurokinin-1 antagonist (NK1a) inhibition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No